CLINICAL TRIAL: NCT02134639
Title: Development of an Innovative Gallium 68 Radiolabeling of DOTATOC (68Ga-DOTATOC) for PET-CT Imaging of Neuro-endocrine Tumors and Preliminary Clinical Evaluation
Brief Title: PET-CT Imaging of Neuro-endocrine Tumors and Preliminary Clinical Evaluation
Acronym: GALTEP
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX2012/28; 2013-003927-12 (EudraCT Number)
Record Dates: First submitted 2014-02-04; First posted 2014-05-09 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient who is suspected of endocrine tumors: According to symptomatology, biology or imaging or pathological context
  Interventions: Procedure: 68Ga-DOTATOC PET-CT Imaging

INTERVENTIONS:
Procedure: 68Ga-DOTATOC PET-CT Imaging

SUMMARY:
Through the investigators involvement in an international consortium, the investigators had the opportunity to acquire a new type of synthetizer for the radiolabelling of such tracers. The investigators propose in this project to develop on their site, the radiosynthesis of 68Ga-DOTATOC and to evaluate prospectively the diagnosis of neuroendocrine tumors, compared with the current imaging OctreoScan®. The objectives of this project are: - to validate the radiosynthesis of 68Ga-DOTATOC on their site with a new synthetizer - and clinically evaluate, through a prospective preliminary study, the diagnostic accuracy of PET-CT with 68Ga-DOTATOC in comparison with other standard imaging examinations.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Patient who is suspected of endocrine tumors according to symptomatology, biology or imaging or pathological context (multiple endocrine neoplasia type 1)
* initial staging: this includes research multifocal disease or locoregional or metastatic extension if well-differentiated neuroendocrine tumor (grade 1 et/ou 2)
* Search of the primary tumor, especially in the case of the inaugural discovery of metastases
* staging of a known recurrence
* Search occult recurrence or suspicion of recurrence (clinical, laboratory, imaging doubtful)
* Patient who have received in a lower range than 2 months of cervico-thoraco-abdominal-pelvic CT and scintigraphy in OctréoScan®
* Patient who have signed an informed consent
* Patient affiliated or beneficiary of regime of social security of a Member State of the European community

Exclusion Criteria:

* Patient with another evolutive cancer disease and/or treated for less than 5 years
* Pregnant or lactating woman
* Premenopausal woman without effective contraception (estrogen-progestin or intrauterine contraceptive device)
* Patient unable to give their free and informed consent
* Persons placed under judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who is suspected of endocrine tumors
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of PET imaging | Inclusion (day 0)
  The diagnostic performance of PET-CT will be calculated and compared with other standard exams as the gold standard histology and clinical follow-up.

SECONDARY OUTCOMES:
Reproducibility | Inclusion (day 0)
  The reproducibility of the new method of radiolabelling will be evaluated by the number of failed syntheses
Tolerance | Inclusion (day 0) and until end of follow up (day 28)
  Tolerance of the tracer will be assessed by the collection of possible side effects
Impact on the therapeutic management | End of follow up (day 28)
  The impact on the therapeutic management of patients will be studied by the analysis of questionnaires with or without taking into account, the results of the PET-CT with 68Ga-DOTATOC.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe FERNANDEZ, Professor, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France